CLINICAL TRIAL: NCT05592236
Title: Effects of Dynamic Compression Garments on Posture, Trunk Control and Upper Extremity Functions in Children With Hemiparetic CP
Brief Title: Effects of Dynamic Compression Garments in Children With CP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ayse Zengin Alpozgen, Assist. Prof, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 004
Record Dates: First submitted 2022-10-20; First posted 2022-10-24 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; dynamic compression; postural control; trunk control; upper extremity function
MeSH Terms: conditions — Cerebral Palsy | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Dynamic compression garments for 2 hours a day in addition to standard therapy twice a week (1 session of 45 minutes) for a total of 6 weeks
  Interventions: Other: Dynamic compression garments; Other: Standard therapy
- Control Group (Active Comparator): Standard therapy twice a week (1 session of 45 minutes) for a total of 6 weeks
  Interventions: Other: Standard therapy

INTERVENTIONS:
Other: Dynamic compression garments — Dynamic compression garments for 2 hours a day in addition to standard therapy twice a week (1 session of 45 minutes) for a total of 6 weeks
  Arms: Study group
Other: Standard therapy — Standard therapy twice a week (1 session of 45 minutes) for a total of 6 weeks

SUMMARY:
In recent years, it is seen that dynamic compression garments are used to increase body stability and to provide tone regulation. Dynamic compression garments are used to apply pressure to specific muscles or muscle groups. Different studies have drawn attention to the effect of dynamic compression garments on postural control and proximal stability. Researchers observed that upper extremity functions and fine motor skills improved with the use of clothing, and they associated this with improved proximal stability. In light of this information, the aim of this study is; To investigate the effects of dynamic compression garments applied in addition to traditional treatment on posture, trunk control, and upper extremity functions during sitting in children with hemiparetic CP.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a group of permanent neurodevelopmental disorders in the development of movement and posture, non-progressive, resulting in activity limitations, resulting from an injury to the developing brain. Children with CP who have problems in sensorimotor coordination due to decreased muscle strength and impaired sensory processing experience postural control problems. In hemiparetic CP, deterioration in the upper extremities affects children's daily living activities such as eating, dressing, undressing, combing hair, brushing teeth, self-care skills, functional independence, and quality of life. Since the trunk plays a very important role in postural control and extremity functions, providing trunk stability and thus effective use of the extremities is one of the important goals of physiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Being diagnosed with congenital spastic hemiparetic cerebral palsy,
2. To be between the ages of 4-18
3. To be at the level of I, II or III according to the Manual Ability Classification System
4. Having sufficient communication skills
5. The willingness of the family and the child to be included in the study

Exclusion Criteria:

1. The family's refusal to participate in the study
2. Botulinum toxin application to the upper extremity or having undergone upper extremity surgery in the last 6 months
3. Having behavioral and communication problems that hinder the practices to be carried out within the scope of the study
4. Having an epileptic seizure

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-06-15 (Estimated); Primary Completion 2023-11-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Manual Ability Classification System | 8 weeks
  Individuals' manual dexterity will be classified according to Manual Ability Classification System before treatment. Manual Ability Classification System is a 5-level classification system developed to classify how children with cerebral palsy aged 4-18 use their hands while holding objects during activities of daily living.
Sitting Assessment Scale | 8 weeks
  It is a standard video-based observation tool designed for the assessment of sitting in children with cerebra palsy. The scale consists of five items: head control, trunk control, foot control, arm functions and hand functions and is evaluated as follows: 1= none; 2= weak; 3= reasonable; 4 = good. Minimum and maximum scores range from 5 to 20.
The Trunk Control Measurement Scale | 8 weeks
  The Trunk Control Measurement Scale measures two key components of trunk control during functional activities. For this reason, the scale consists of two parts: Static Sitting Balance and Dynamic Sitting Balance. The scale consists of 15 items in total. While the total score of the scale varies between 0-58 points, higher scores indicate a better performance.
Quality of Upper Extremity Skills Test | 8 weeks
  It is a test that evaluates the quality of movement and manual skills of children with cerebral palsy. It deals with how the child does the activity. It consists of 7 parts. The evaluator scores the test by observing how the child performs the desired movements. The increase in the score obtained from the test indicates the increase in the quality of upper extremity skills.
ABILHAND-Kids: a measure of manual ability | 8 weeks
  ABILHAND-Kids is a 21-item scale that evaluates bilateral hand use in activities of daily living in children with cerebral palsy. Each sub-item evaluates the difficulty level of children while performing the activity at three levels as impossible, difficult and easy.
Shriners Hospital Upper Extremity Evaluation | 8 weeks
  It is an upper extremity movement and function assessment tool based on video observation for children aged 3-18 years. It consists of 3 sub-sections: positional dynamic analysis, spontaneous functional analysis and catch-release function.
The Pediatric Evaluation of Disability Inventory | 8 weeks
  It is a scale used to evaluate changes in performance, functional skills and functional skills in children. It consists of 3 subsections. These; "Functional skills", "Caregiver level of help" and "Adaptations". Each division consists of the areas of self-care, mobility and social function. Functional skills subsection will be used in accordance with the purpose of our study.